CLINICAL TRIAL: NCT03959397
Title: A Real-world Study of Paclitaxel Injection (Albumin-bound) for Neoadjuvant Treatment of Breast Cancer
Brief Title: Paclitaxel Injection (Albumin-bound) for Neoadjuvant Treatment of Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Aiping shi, Chief physician and associate professor, Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-KAL-BC-12
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer Stage
Keywords: Breast cancer; neoadjuvant therapy; Nab-paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nab-paclitaxel (Experimental): nab-paclitaxel monotherapy or combination therapeutic regimen
  Interventions: Drug: nab-paclitaxel

INTERVENTIONS:
Drug: nab-paclitaxel — nab-paclitaxel monotherapy or combination therapeutic regimen
  Other Names: ABRAXANE ，Albumin-binding paclitaxel

SUMMARY:
Neoadjuvant chemotherapy is a systemic cytotoxic drug therapy for non-metastatic tumors before local therapy, Now it has become an important part of standard treatment for a stage II, III, and the first clinical Ⅳ breast cancer .Both domestic and foreign authoritative guidelines recommend the use of albumin-binding paclitaxel in the neoadjuvant treatment of breast cancer .In addition, clinical studies at home and abroad have preliminarily confirmed the application value and therapeutic benefit of albumin-binding paclitaxel in breast cancer neoadjuvant therapy, and the toxic and side effects can be tolerated.

DETAILED DESCRIPTION:
Data were collected on the efficacy and safety of neoadjuvant therapy in patients receiving albumin-binding taxol regimens,Subgroup analysis was performed for different treatment regimens, dosages, molecular subtypes and tumor stages,To further screen the dominant population and the chemotherapy regimen with clinical benefit of albumin paclitaxel, so as to provide evidence-based medical evidence for breast cancer neoadjuvant clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed content obtained prior to treatment. The patients were fully explained and understood the purpose, contents, predicted efficacy, pharmacological effects, and risks of this study.
2. target population 1)The histologic diagnosis of the primary invasive breast cancer and clinical stage I - III, first option Ⅳ period; 2) One of the following conditions:Large mass (>3cm);Axillary lymph node metastasis;her-2 positive; tri-negative; For those who are willing to preserve breast, but have difficulty in breast conserving due to the large proportion of tumor size and breast volume; 3) The clinician determined that the patient was suitable for the treatment with albumin-binding taxol regimen;4) The subjects have good compliance, can be treated and followed up, and voluntarily comply with the relevant provisions of this study 5)No contraindications for nab-paclitaxel.
3. Age and reproductive status 1) Age ≥ 18 years 2) Subjects of child-bearing age must agree to take effective contraceptive measures during the study period; Serum or urine pregnancy tests must be negative for women of childbearing age 24 hours before the start of chemotherapy; 3) Women must not lactate.

Exclusion Criteria:

1. Allergy to paclitaxel for injection (albumin binding) and/or its adjuvants has been demonstrated;
2. Pregnant or lactating women
3. Abnormal results of physical examination and laboratory examination 1) Absolute neutrophil count (ANC) 90g/L 1.5 × 109/L; Platelets (PLT) 90g/L 100 × 109/L; Hemoglobin (Hgb) < 90g/L 2) Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/ alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) >2.5 × institutional upper limit of normal (ULN), >5 × institutional upper limit of normal (ULN) (hepatic metastases); Total bilirubin (TBIL)>1.5 × ULN; 3) Creatinine (CRE)> 1.5 × ULN 4) Prothrombin time (PT) and international normalized ratio (INR) > 1.5 × ULN. Unless the subject had received anticoagulant treatment
4. Paclitaxel for injection (albumin binding type) contraindications in patients
5. Participating in clinical trials of other taxoids
6. Patients with concomitant other tumors, other than cured carcinoma in situ of the cervix and non-melanoma skin cancer
7. Participation in any trial drug treatment or another interventional clinical trial 30 days before screening period.
8. The researchers considered that there were other conditions that were not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
the Pathological complete remission(pCR) | 2 weeks
  Histopathological examination of breast and axillary lymph node specimens without invasive cancer cell remnants. Complete pathological response is also considered to be achieved if only in situ cancer cell remnants are present in the surgical specimens.
Disease-free survival (DFS) | 6 months
  defined as the time from the beginning of randomization to recurrence or death due to disease progression

SECONDARY OUTCOMES:
the overall survival (OS) | 6 months
  defined as the time between enrollment in the study (i.e., ICF) and death from any cause.Subjects who survived the last contact were deleted on the last contact date
Breast conserving rate | 6 months
  after neoadjuvant treatment, the percentage of patients undergoing breast conserving surgery in the total number of evaluable cases.

OTHER OUTCOMES:
Adverse events (AE) | 6 months
  Adverse events (AE) were monitored on an ongoing basis and classified according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Fan zhimin, Doctor, Study Director — The First Hospital of Jilin University
Locations (1):
- the first hospital of Jilin University, Jilin, Changchun, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Untch M, Jackisch C, Schneeweiss A, Conrad B, Aktas B, Denkert C, Eidtmann H, Wiebringhaus H, Kummel S, Hilfrich J, Warm M, Paepke S, Just M, Hanusch C, Hackmann J, Blohmer JU, Clemens M, Darb-Esfahani S, Schmitt WD, Dan Costa S, Gerber B, Engels K, Nekljudova V, Loibl S, von Minckwitz G; German Breast Group (GBG); Arbeitsgemeinschaft Gynakologische Onkologie-Breast (AGO-B) Investigators. Nab-paclitaxel versus solvent-based paclitaxel in neoadjuvant chemotherapy for early breast cancer (GeparSepto-GBG 69): a randomised, phase 3 trial. Lancet Oncol. 2016 Mar;17(3):345-356. doi: 10.1016/S1470-2045(15)00542-2. Epub 2016 Feb 8. PMID 26869049
- [Background] Gluz O, Nitz U, Liedtke C, Christgen M, Grischke EM, Forstbauer H, Braun M, Warm M, Hackmann J, Uleer C, Aktas B, Schumacher C, Bangemann N, Lindner C, Kuemmel S, Clemens M, Potenberg J, Staib P, Kohls A, von Schumann R, Kates R, Kates R, Schumacher J, Wuerstlein R, Kreipe HH, Harbeck N. Comparison of Neoadjuvant Nab-Paclitaxel+Carboplatin vs Nab-Paclitaxel+Gemcitabine in Triple-Negative Breast Cancer: Randomized WSG-ADAPT-TN Trial Results. J Natl Cancer Inst. 2018 Jun 1;110(6):628-637. doi: 10.1093/jnci/djx258. PMID 29228315
- [Background] Zong Y, Wu J, Shen K. Nanoparticle albumin-bound paclitaxel as neoadjuvant chemotherapy of breast cancer: a systematic review and meta-analysis. Oncotarget. 2017 Mar 7;8(10):17360-17372. doi: 10.18632/oncotarget.14477. PMID 28061451
- [Background] Nahleh ZA, Barlow WE, Hayes DF, Schott AF, Gralow JR, Sikov WM, Perez EA, Chennuru S, Mirshahidi HR, Corso SW, Lew DL, Pusztai L, Livingston RB, Hortobagyi GN. SWOG S0800 (NCI CDR0000636131): addition of bevacizumab to neoadjuvant nab-paclitaxel with dose-dense doxorubicin and cyclophosphamide improves pathologic complete response (pCR) rates in inflammatory or locally advanced breast cancer. Breast Cancer Res Treat. 2016 Aug;158(3):485-95. doi: 10.1007/s10549-016-3889-6. Epub 2016 Jul 8. PMID 27393622